CLINICAL TRIAL: NCT06572397
Title: An Open-Label Study Assessing the Ocular and Systemic Safety and Systemic Absorption of H1337 Ophthalmic Solution, 1% in Healthy Volunteers
Brief Title: Open-Label Study of Safety of H1337 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: D. Western Therapeutics Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H1337-CS101
Record Dates: First submitted 2024-08-22; First posted 2024-08-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-10

CONDITIONS: Glaucoma Open-Angle Primary; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- H-1337 1.0% Ophthalmic Solution b.i.d. (Experimental): One drop H-1337 twice daily in the both eyes for 7 days
  Interventions: Drug: H-1337 1.0%

INTERVENTIONS:
Drug: H-1337 1.0% — ophthalmic solution

SUMMARY:
The trial will evaluate the safety of one dose regimen of H-1337 [1% twice daily (b.i.d.)] in both eyes in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female subjects
* Subjects in good ocular and systemic health with clinically insignificant medical and ophthalmic history

Exclusion Criteria:

* Chronic or acute ophthalmic disease in each eye including but not limited to any form of glaucoma, retinal diseases, clinically significant cataract (primary or secondary)
* Recent intraocular surgery in either eye (within 6 months)

Note: Other inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events Reporting [Safety and Tolerability] | Screening through Day 9
  Incidence of ocular and systemic adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Research Foundation Inc., Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No